CLINICAL TRIAL: NCT03088267
Title: Dyanavel® XR Extended-Release Oral Suspension in the Treatment of Children Wit
Brief Title: Dyanavel® XR Extended-Release Oral Suspension in the Treatment of Children With ADHD: A Laboratory School Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRI102-ADD-300
Record Dates: First submitted 2017-03-09; First posted 2017-03-23 (Actual); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, two treatment, two sequence, placebo-controlled crossover study
Who Masked: Participant, Investigator
Masking Description: placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment (Active Comparator): Double blind amphetamine extended-release oral suspension, 2.5 mg/mL, 6, 7 or 8 mL po QAM
  Interventions: Drug: amphetamine extended-release oral suspension, 2.5 mg/mL; Drug: Placebo extended-release oral suspension
- Placebo Treatment (Placebo Comparator): Double blind placebo, 6, 7 or 8 mL po QAM
  Interventions: Drug: amphetamine extended-release oral suspension, 2.5 mg/mL; Drug: Placebo extended-release oral suspension

INTERVENTIONS:
Drug: amphetamine extended-release oral suspension, 2.5 mg/mL — 5 mL1 (5 mg), 7 mL (17.5 mg) or 8 mL (20 mg) PO
  Other Names: Dyanavel XR
Drug: Placebo extended-release oral suspension — 6, 7 or 8 mL PO

SUMMARY:
This study was conducted to assess the efficacy and safety of DYANAVEL XR (amphetamine extended-release oral suspension, CII) for the treatment of symptoms of attention-deficit/hyperactivity disorder (ADHD) in children aged 6-12 years.

DETAILED DESCRIPTION:
This is a randomized, double-blind, two treatment, two sequence, placebo-controlled crossover study to assess the efficacy and safety of dose Dyanavel XR in reducing signs and symptoms of ADHD compared with placebo in pediatric subjects ages 6 to 12 years with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 6 to 12 years at the time of screening, inclusive
2. Diagnosed with ADHD by a psychiatrist within 6 months of study enrolment or newly diagnosed with ADHD using the DSM-5 criteria for ADHD
3. An ADHD-RS-5 score at Screening ≥90th percentile for sex and age in at least one of the following categories:

   1. Hyperactive-impulsive subscale,
   2. Inattentive subscale, or
   3. Total score. Subjects who do not meet this criteria at screening can have ADHD-RS-5 repeated at baseline, after washout of stimulant medication for a minimum of 24 hours prior to baseline.
4. In the clinical judgment of the Investigator, the subject must be in need of pharmacological treatment for ADHD.
5. Females of childbearing potential must be non-lactating and must have a negative serum pregnancy test at screening
6. Provide written informed consent (parent/guardian) and assent (child aged 10 - 12 years only) prior to participation in the study

Exclusion Criteria:

1. Diagnosed with any DSM-5 active disorder (other than ADHD) with the exception of specific phobias, learning disorders, motor skills disorders, communication disorders, oppositional defiant disorder, elimination disorders, and sleep disorders
2. Known history of chronic medical illnesses including severe hypertension, untreated thyroid disease, peripheral vasculopathy, known structural cardiac disorders, serious cardiac conditions, serious arrhythmias, cardiomyopathy, known family history of sudden death
3. Known history or presence of significant renal or hepatic disease, as indicated by clinical laboratory assessment (liver function test results ≥ two times the upper limit of normal, blood urea nitrogen, or creatinine).
4. Clinically significant abnormal ECG or cardiac findings on physical examination (including the presence of a pathologic murmur)
5. Use of the following medications within 30 days of Baseline Visit:

   * MAOI - monoamine oxidase inhibitors (e.g., Selegiline, isocarboxazid, phenelzine, tranylcypromine)
   * Tricyclic Antidepressants (e.g. Desipramine, protriptyline)
6. Use of the following medications within 3 days of Baseline Visit

   * Gastrointestinal acidifying agents (e.g., guanethidine, reserpine, glutamic acid HCl, ascorbic acid)
   * Urinary acidifying agents (e.g., ammonium chloride, sodium acid phosphate, methenamine salts)
7. Use of atomoxetine within 14 days of Baseline Visit
8. Planned use of prohibited drugs or agents from the Screening visit through the end of the study
9. Abnormal clinically significantly laboratory test value at screening that, in the opinion of the Investigator, would preclude study participation
10. Known history of allergy/hypersensitivity to amphetamine or any of the components of Dyanavel XR, or topical anaesthetics
11. Known history of lack of response to amphetamine
12. Parent or guardian's inability or unwillingness to follow directions of the Investigator or study research staff.
13. Any uncontrolled medical condition that in the opinion of the Investigator would preclude study participation
14. History of significant illness requiring hospitalization, or surgery requiring anaesthetics within 30 days of Baseline Visit

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2017-02-25 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Berry, MD, PhD, Study Chair — Tris Pharma
Locations (1):
- Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Childress AC, Kando JC, King TR, Pardo A, Herman BK. Early-Onset Efficacy and Safety Pilot Study of Amphetamine Extended-Release Oral Suspension in the Treatment of Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2019 Feb;29(1):2-8. doi: 10.1089/cap.2018.0078. Epub 2018 Dec 21. PMID 30575407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date first subject enrolled: February 11, 2017 Date last subject completed: February 25, 2017
Pre-assignment Details: All 18 subjects were enrolled and completed the study.
Groups:
- Sequence: AMPH EROS/Placebo: Patients optimized on open label dose of AMPH EROS. Randomized to optimized dose of AMPH EROS for 1 day. Laboratory classroom assessment takes place. Then crossover to placebo for 4-5 days followed by second laboratory classroom assessment.
- Sequence: Placebo/AMPH EROS: Patients optimized on open label dose of AMPH EROS. Randomized to placebo for 1 day. Laboratory classroom assessment takes place. Then crossover to optimized dose of AMPH EROS for 4-5 days followed by second laboratory classroom assessment.
Period: Overall Study
Arm/Group | Sequence: AMPH EROS/Placebo | Sequence: Placebo/AMPH EROS
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Open label phase: amphetamine extended-release oral suspension, 2.5 mg/mL at optimal dose
  Double blind phase:
  A single dose of amphetamine extended-release oral suspension, 2.5 mg/mL, 6, 7 or 8 mL po QAM, or placebo extended-release oral suspension: 6, 7 or 8 mL PO
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Age, Customized [Median (Full Range); unit: years] | 10 [6 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Combined Scores, Baseline to 30 Minutes Post Dose
Description: Change in SKAMP-C (Swanson, Kotkin, Agler, M-Flynn, and Pelham combined) score from pre-dose, by treatment. The SKAMP-C is a rating scale that assesses functional impairment related to ADHD in the classroom, including the performance of academic tasks, following class rules, and interacting with peers and adults in the classroom. The SKAMP-C is a 13-item, 7-score rating system (0=normal to 7=maximal impairment). The higher the score, the worse the impairment. A decrease from baseline in the combined (all 13 items) score indicates improvement. The SKAMP-C is used to assess the time course of treatment effects in laboratory classroom studies.
Time Frame: Change in SKAMP-C score from baseline to 30 minutes postdose.
Population: Intent to Treat Population: 18 subjects
Measure: Least Squares Mean (Standard Error); unit: number of questions answered correctly
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 18 | 18
number of questions answered correctly | -6.1 (2.29) | 2.5 (2.29)
Statistical Analysis 1: Comparison: Active Treatment vs Placebo Treatment; Test type: Superiority; p = 0.0118, ANCOVA; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-14.94 to -2.17]

2. Secondary Outcome: Change in Permanent Product Measure of Performance (PERMP-C) Score (Problems Answered Correctly)
Description: Change from pre-dose in PERMP-C scores (Permanent Product Measure of Performance; defined as the number of problems attempted and number of problems solved correctly) at 30 minutes post-dose and at 3 hours post-dose. The PERMP-C is designed to assess compliance and academic productivity in school children. It is a 10-minute timed test in which the number of problems attempted and correct are assessed prior to and after an intervention. Scoring is based on problems attempted and correct. An increase in numerical score is indicative of improvement.
Time Frame: 30 minutes postdose and 3 hours postdose
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: Change from baseline in PERMP score
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 18 | 18
Change from baseline in PERMP score
  Change from predose in PERMP-C at 30 minutes | 14.4 (7.25) | -4.7 (7.25)
  Change from predose in PERMP-C at 3 hours | 52.4 (9.43) | -7.9 (9.43)
Statistical Analysis 1: Comparison: Active Treatment vs Placebo Treatment; Comparison at 30 minutes post-dose; Test type: Superiority; p = 0.1128, ANCOVA; Mean Difference (Final Values) = 18.8, 95% CI 2-sided [-4.94 to 42.50]
Statistical Analysis 2: Comparison: Active Treatment vs Placebo Treatment; Comparison at 3 hours postdose; Test type: Superiority; p = 0.0003, ANCOVA; Mean Difference (Final Values) = 60.3, 95% CI 2-sided [32.91 to 87.75]

ADVERSE EVENTS:
Time Frame: The duration of the study (5 weeks from screening to final follow-up assessment)
Groups:
- AMPH EROS: Open Label Phase: All AEs reported are from the open-label dose optimization phase with AMPH EROS. The open-label dose optimization phase preceded the crossover portion of the study.
- Crossover Phase: AMPH EROS; Crossover Phase: Placebo: These AEs occurred during the crossover phase of the study.
Arm/Group | AMPH EROS: Open Label Phase | Crossover Phase: AMPH EROS | Crossover Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 6/18 | 0/18 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMPH EROS: Open Label Phase (N=18) | Crossover Phase: AMPH EROS (N=18) | Crossover Phase: Placebo (N=18)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | NA | NA
Bronchitis (Infections and infestations) | 1 (1) | NA | NA
Respiratory tract viral infection (Infections and infestations) | 1 (1) | NA | NA
Abdominal pain, upper (Gastrointestinal disorders) | 2 (2) | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA | NA
Fatigue (General disorders) | 3 (3) | NA | NA
Headache (Nervous system disorders) | 2 (2) | NA | NA
Motion sickness (Nervous system disorders) | 1 (1) | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | NA | NA
Affect lability (Psychiatric disorders) | 2 (2) | NA | NA
Constricted affect (Psychiatric disorders) | 1 (1) | NA | NA
Visioned blurred (Eye disorders) | 1 (1) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03088267/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03088267/SAP_001.pdf